CLINICAL TRIAL: NCT02340065
Title: Endocuff-assisted vs. Standard Colonoscopy: a Randomized, Back-to-Back Study
Brief Title: Endocuff-assisted vs. Standard Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, ATHANASIOS SIOULAS, Dr, Attikon Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: ENDOCUFF-001
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Colon Neoplasms
Keywords: colonoscopy; adenoma detection rate; Endocuff-assisted colonoscopy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard colonoscopy (Active Comparator): total polyp/adenoma detection with standard colonoscopy, polyp/adenoma detection in the right colon with standard colonoscopy
  Interventions: Procedure: Endocuff-assisted colonoscopy
- Endocuff-assisted colonoscopy (Active Comparator): total polyp/adenoma detection with Endocuff-assisted colonoscopy, polyp/adenoma detection in the right colon with Endocuff-assisted colonoscopy
  Interventions: Procedure: standard colonoscopy

INTERVENTIONS:
Procedure: standard colonoscopy — examination of the colon with a conventional colonoscope
  Other Names: conventional colonoscopy
  Arms: Endocuff-assisted colonoscopy
Procedure: Endocuff-assisted colonoscopy — examination of the colon with Endocuff-assisted colonoscopy
  Other Names: Endocuff
  Arms: standard colonoscopy

SUMMARY:
The aim of this study is to evaluate Endocuff- assisted colonoscopy in terms of its possible additive contribution in the detection of important lesions, namely polyps and cancers, compared to standard colonoscopy, in a series of patients undergoing back-to-back screening or surveillance colonoscopies in a randomized fashion. Moreover, we aim to assess possible changes regarding post-polypectomy surveillance programs following Endocuff utilization.

DETAILED DESCRIPTION:
Tandem colonoscopies studies results, show that novel endoscopic technologies detect about 20% more adenomas than those conventional colonoscopy does (missed adenomas). Since Endocuff-assisted colonoscopy cannot be considered as a perfect examination, we hypothesize that conventional colonoscopy will detect one third of the missed adenomas that Endocuff-assisted colonoscopy detects in a similar setting. Therefore a sample size of 120 adenomas achieves 80% power to detect an odds ratio of 3.0 using a two-sided McNemar test with a significance level of 0.05. The odds ratio is equivalent to a difference between two paired proportions of 14% which occurs when the proportion of detected missed adenomas during Endocuff-assisted colonoscopy is 21% and the proportion of missed adenomas during conventional colonoscopy is 7%. During one year period before the study initiation, our colonoscopy performance quality data show that we detect a mean number of adenomas per patient equal of 0.7 in a population similar to the one recruited in our study. Therefore, 172 patients overall will be required to detect 120 adenomas. Given the uncertainty of our estimation and in order to cope with patients exclusions, withdrawals and unexpected incomplete colonoscopies, we decided to recruit 200 patients.

A more extensive description regarding the investigators study is provided in the following fields.

ELIGIBILITY:
Inclusion Criteria:

* adults undergoing elective screening or surveillance colonoscopy
* symptomatic adults with indication for colonoscopy

Exclusion Criteria:

* age<18 and > 80 years
* poor overall health (ASA III, IV)
* recent abdominal surgery
* presence of abdominal wall hernias
* active colitis
* previous bowel resection
* inflammatory bowel disease
* polyposis syndromes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
number and rate of missed adenomas | one week
  in the entire colon

SECONDARY OUTCOMES:
number of adenomas and adenoma detection rate in the entire colon | one week
  with both Endocuff-assisted and standard colonoscopy
number of adenomas and adenoma detection rate in the right colon | one week
  with both Endocuff-assisted and standard colonoscopy
number of polyps and polyp detection rate in the entire colon | one week
  with both Endocuff-assisted and standard colonoscopy
number of polyps and polyp detection rate in the right colon | one week
  with both Endocuff-assisted and standard colonoscopy
colonoscopy completion (colonoscopy completion rate, reason for incomplete colonoscopy) | one week
  colonoscopy completion rate, reason for incomplete colonoscopy
intubation and withdrawal time | one week
  for both Endocuff-assisted and standard colonoscopy (time spent for therapeutic procedures is excluded)
adverse events | one week
  adverse event rate
endoscopist's satisfaction (quantified using a scale from 0 (not satisfied) to 10 (completely satisfied) | one week
  endoscopist's satisfaction quantified using a scale from 0 (not satisfied) to 10 (completely satisfied) for Endocuff-assisted colonoscopy
mean number of adenomas per procedure | one week
  with both Endocuff-assisted and standard colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: KONSTANTINOS TRIANTAFYLLOU, PROF, Study Chair — Hepatogastroenterology Unit, 2nd Department of Internal Medicine and Research Institute, Attikon University General Hospital, University of Athens, Greece; DIMITRIOS POLYMEROS, MD, Study Director — Hepatogastroenterology Unit, 2nd Department of Internal Medicine and Research Institute, Attikon University General Hospital, University of Athens, Greece
Locations (1):
- Hepatogastroenterology Unit, 2nd Department of Internal Medicine and Research Institute, Attikon University General Hospital, Haidari, Attica, Greece

REFERENCES:
- [Background] Floer M, Biecker E, Fitzlaff R, Roming H, Ameis D, Heinecke A, Kunsch S, Ellenrieder V, Strobel P, Schepke M, Meister T. Higher adenoma detection rates with endocuff-assisted colonoscopy - a randomized controlled multicenter trial. PLoS One. 2014 Dec 3;9(12):e114267. doi: 10.1371/journal.pone.0114267. eCollection 2014. PMID 25470133
- [Background] Biecker E, Floer M, Heinecke A, Strobel P, Bohme R, Schepke M, Meister T. Novel endocuff-assisted colonoscopy significantly increases the polyp detection rate: a randomized controlled trial. J Clin Gastroenterol. 2015 May-Jun;49(5):413-8. doi: 10.1097/MCG.0000000000000166. PMID 24921209
- [Derived] Triantafyllou K, Polymeros D, Apostolopoulos P, Lopes Brandao C, Gkolfakis P, Repici A, Papanikolaou IS, Dinis-Ribeiro M, Alexandrakis G, Hassan C. Endocuff-assisted colonoscopy is associated with a lower adenoma miss rate: a multicenter randomized tandem study. Endoscopy. 2017 Nov;49(11):1051-1060. doi: 10.1055/s-0043-114412. Epub 2017 Aug 1. PMID 28763808